CLINICAL TRIAL: NCT02342002
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Missed Abortion: A Randomized-controlled Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1015
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-11

CONDITIONS: Missed Abortion; Pregnancy
Keywords: mifepristone; misoprostol; obstetrics; reproductive health; pregnancy; abortion; missed abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone-misoprostol regimen (Experimental): After a woman is determined eligible and signs the informed consent document, she will receive 200 mg mifepristone and advised to swallow the pill when they arrive at home. 24 hours after administration of the mifepristone, women will administer the four tablets of 200 mcg misoprostol sublingually.
  Interventions: Drug: Mifepristone; Drug: Misoprostol
- Misoprostol alone regimen (Placebo Comparator): After a woman is determined eligible and signs the informed consent document, she will receive a placebo (of same shape and size of mifepristone) and advised to swallow the pill when they arrive at home. 24 hours after administration of the mifepristone, women will administer the four tablets of 200 mcg misoprostol sublingually.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Mifepristone for treatment of missed abortion
  Arms: Mifepristone-misoprostol regimen
Drug: Misoprostol — Misoprostol for treatment of missed abortion

SUMMARY:
The purpose of the proposed study is to compare - in a randomized, placebo-controlled, double-blinded trial - a combination of mifepristone and misoprostol to misoprostol used alone for missed abortion.

DETAILED DESCRIPTION:
The primary aim of this trial is to compare the efficacy of mifepristone-misoprostol versus misoprostol alone for treatment of missed abortion. This will be a randomized controlled double-blinded trial of 416 women comparing misoprostol alone to mifepristone plus misoprostol for treatment of missed abortion less than 13 weeks+ 0 days LMP. All women in the trial will undergo routine screening (including ultrasound) and pre-medical induction care per standard practice at the hospital. All eligible women agreeing to participate in the study will be randomized to receive one of the following regimens: 1) STUDY GROUP ONE: 200mg mifepristone followed in 24 hours by 800mcg sublingual misoprostol; 2) STUDY GROUP TWO: placebo followed in 24 hours by 800mcg sublingual misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound examination demonstrating:

  1. Evidence of fetal demise (no fetal cardiac activity despite recognizable embryo and dates consistent with the likelihood of visible pregnancy) OR
  2. Empty gestational sac with no evidence of incomplete abortion or growth over a 7-day period confirmed by two ultrasounds performed one week apart.
* If fetus exists, fetal size less than 12 weeks+6 days
* Closed cervical os
* Eligible to consent for research according to local regulations

Exclusion Criteria:

* Active bleeding at enrollment and/or history of bleeding within the prior week
* Allergies or other contraindications to the use of mifepristone or misoprostol
* Suspected ectopic pregnancy
* History of trophoblastic disease
* Coagulation disorder and/or currently taking anticoagulants
* Any serious medical condition

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 416 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of successful evacuation of the uterus | 1 week after treatment
  uterine evacuation without the need for uterine aspiration or other surgery

SECONDARY OUTCOMES:
Rate of successful evacuation without any additional intervention | 1 week after treatment
  uterine evacuation without the need for vacuum aspiration, additional uterotonics or other intervention
Excessive bleeding or a complication for which a woman received treatment | 30 days after treatment
Induction expulsion interval after misoprostol administration | one week follow-up
  time interval between misoprostol administration and the expulsion
Acceptability of assigned method to women | one week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Principal Investigator — Gynuity Health Projects
Locations (4):
- Hospital Nacional Profesor Alejandro Posadas, Buenos Aires, Argentina
- CHU Libreville, Libreville, Gabon
- Hospital General Valle Ceylan, Tlalnepantla, Mexico
- Agha Khan University Hospital, Karachi, Pakistan